CLINICAL TRIAL: NCT05656612
Title: The Effect of Education Given at Different Times Before a Breast Biopsy on Anxiety, Readiness for the Procedure, Satisfaction, and Pain Levels in Women: A Randomized Study
Brief Title: The Effect of Education Given at Different Times Before a Breast Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Cansu Cil, specialist nurse, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Breast Biopsy
Record Dates: First submitted 2022-09-30; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Educational Problems; Bypass Complication
Keywords: breast biopsy; anxiety; pain; satisfaction; patient education; nursing
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Group Given Training 1-2 Weeks Before The Procedure (Experimental): Participants received breast biopsy procedure training once. 1-2 weeks before the breast biopsy procedure.
  Interventions: Other: Written, Oral and Visual Education
- The group trained on the day of the procedure (Experimental): Participants received one time breast biopsy procedure training. The day of the breast biopsy procedure.
  Interventions: Other: Written, Oral and Visual Education
- Repetitive training group (Experimental): Participants received twice breast biopsy procedure training. The first training is 1-2 weeks before the breast biopsy procedure. The second training is the day of the breast biopsy procedure.
  Interventions: Other: Written, Oral and Visual Education

INTERVENTIONS:
Other: Written, Oral and Visual Education — Before the training, state anxiety levels were measured with a questionnaire. The pre-process measurement was repeated. Post-procedure pain and satisfaction levels were measured using a scale.
  Arms: The Group Given Training 1-2 Weeks Before The Procedure
Other: Written, Oral and Visual Education — Before the training, state anxiety levels were measured with a questionnaire. The pre-process measurement was repeated. Post-procedure pain and satisfaction levels were measured using a scale.
  Arms: The group trained on the day of the procedure
Other: Written, Oral and Visual Education — Before the initial training was given, state anxiety levels were measured with a questionnaire.
  The pre-process measurement was repeated. Post-procedure pain and satisfaction levels were measured using a scale.
  Arms: Repetitive training group

SUMMARY:
Aim: This study was conducted to investigate the effect of education given at different times before a breast biopsy on anxiety, readiness for the procedure, pain, and satisfaction levels in women. Background: A breast biopsy is an invasive procedure that causes pain and anxiety. Patient education is an effective and evidence-based nursing intervention that reduces pain and anxiety levels. Design: The study is a single-center, uncontrolled randomized clinical trial. Method: Participants (n: 60) in the study were randomly assigned into three groups. The first group (n: 20) was given education about the breast biopsy 1-2 weeks before the procedure, the second group (n: 20) was given education on the day of the procedure, and the third group (n: 20) was given education at two different times, the first 1-2 weeks before the procedure and the second on the day of the procedure. Research data were collected by using a Descriptive Characteristics Form, the State Anxiety Inventory, and a Patient Assessment Form.

DETAILED DESCRIPTION:
INTRODUCTION Breast cancer has the highest incidence among women worldwide. Of the three methods (physical examination, imaging, and biopsy) in the diagnosis of breast lesions and breast cancer, the biopsy is a frequently used standard. A breast biopsy is a safe and effective diagnostic method, but it causes pain and anxiety, especially for those who will have a biopsy for the first time. Considering the clinically significant anxiety levels experienced by women before a biopsy, it is necessary to develop strategies to help them manage their anxiety better. Various studies have shown that uncertainty about the biopsy procedure is associated with high levels of anxiety, and women experience less anxiety and other negative emotions if they are given reassuring information about the procedure. However, no study has been found in the literature regarding the optimal time for patient education to be planned for a breast biopsy. There is a need to determine the most accurate time for patient education. Although there are many studies on education methods to reduce anxiety and other related problems before interventional procedures, the optimal time for this education is still being debated. It is considered that there is a need for research into determining the most effective education time for patient education to be given before a breast biopsy.

RESEARCH QUESTION AND OBJECTIVES Although the effectiveness of educational interventions in reducing the anxiety and pain levels of patients and increasing their readiness and satisfaction for the procedure before a breast biopsy has been shown, very little is known about the optimal time for this educational intervention. Knowledge of the optimal education time will both increase patient comfort in the best way and help us to manage the personnel workforce and cost in the best way. Therefore, this study was conducted to evaluate the effects of patient education given at different times before a breast biopsy on anxiety, readiness for the procedure, pain, and satisfaction levels in women.

Hypotheses of the Research:

H0: There is no difference between patients who receive education 1-2 weeks before a breast biopsy, patients who receive education on the day of the procedure, and patients who receive repetitive education at both times in terms of anxiety, readiness, pain, and satisfaction levels.

H1: There is a difference between patients who receive education 1-2 weeks before a breast biopsy, patients who receive education on the day of the procedure, and patients who receive repetitive education at both times in terms of anxiety, readiness, pain, and satisfaction levels.

METHOD

Study design:

This is a single-center, randomized clinical trial. It was conducted in the radiology clinic of a training and research hospital between August 2020 and October 2020. This article follows the requirements of CONSORT statement.

Ethical aspects:

At the outset, the permission of the Non-Interventional Research Ethics Committee (decision no: 2020-01/515) and the hospital where the research was conducted was obtained. Patients who met the inclusion criteria were informed about the scope of the study. Verbal and written consent was obtained from the participants.

Participants:

The study sample consisted of women who presented to the aforementioned hospital between August 2020 and October 2020 for a breast biopsy appointment. The sample size was calculated as a total of 54 patients in three groups, based on a 95% confidence interval (1-α), 95% test power (1-β), and an effect size of d=0.826 by considering the mean anxiety values before and after the application in each group according to a similar study. Assuming a 10% loss, the final minimum sample size in the 3 groups was calculated as 60 individuals.

Randomization:

Randomization was made by the researcher by creating a random number sequence in the Microsoft Excel program. The generated random number sequence was divided into 3 research groups and the patients who came to the hospital for the procedure were assigned to the groups according to this list by the researcher.

Blinding:

Patients were informed about the purpose of the study, and all data were collected by the same researcher. Due to the study design, the researcher could not be blinded, but since all participants received education at different times, they did not know which group they were in.

Educational material:

The educational material developed in line with the literature and clinical data was designed as the Breast Biopsy Education Manual and Breast Biopsy Education Video. The content of the education included the definition of breast biopsy, the introduction of the biopsy room, the position of the patient during the procedure, the steps of the procedure, things to consider after the procedure considerations and recommendations, possible risks after the procedure, time to get results, and contact information. The pictures and photographs used in the education booklet and video were prepared by the researcher. Four faculty members in the field of nursing and a specialist in medicine were consulted about the language intelligibility and content of the education.

Implementation of the education program:

The planned patient education was carried out in a room reserved for education. First, participants were given information about the breast biopsy procedure, the education booklet was introduced, and the video, specially prepared for this program, was watched on a personal computer. Patients examined the education booklet. At the same time, patients' questions on the subject were answered by the researcher during the education. The education session took approximately 15 minutes. At the end of the education, patients were told that they could take the booklets home.

The study was carried out in two stages. The first stage was performed when patients came to the radiology clinic to make an appointment for a breast biopsy (approximately 1-2 weeks before the procedure), and the second stage was performed on the day of the procedure.

Stage 1: At this stage, necessary data were collected by the researcher from all the participants by using the data collection forms. The readiness levels of the patients were assessed with the "VAS". Physiological parameters (blood pressure, pulse, and respiratory rate) were measured and recorded with the same device for all patients by the same researcher. All of the participants were routinely informed about what they needed to do before coming to the procedure. After the data collection forms and provision of routine information were completed, the patients were randomized into 3 groups. Women in the first and third groups were given education.

Stage 2: This stage was carried out on the day of the breast biopsy procedure. The women in the second and third groups were given education on the day of the procedure. At this stage, all participants were asked to respond to the State Anxiety Inventory again just before the procedure, and data about the level of readiness and vital signs were recorded before the procedure. After the breast biopsy procedure, data on satisfaction with the procedure, pain, and physiological parameters of all research groups were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women who were older than 18 years of age, had a breast biopsy for the first time, had no communication problems, and volunteered to participate in the study were included in the study.

Exclusion Criteria:

* Women who had major hearing, vision, or speech impairments or those who used antidepressants or anxiolytic drugs were not included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women were studied for the breast biopsy procedure because all patients who come for the procedure are women.
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
initial state anxiety level | It was evaluated 1-2 weeks before the breast biopsy.
  State anxiety levels of patients
change anxiety level | It was evaluated on the day of breast biopsy.
  State anxiety levels of patients
initial readiness level | It was evaluated 1-2 weeks before the day of breast biopsy.
  Patients' level of readiness for the breast biopsy was evaluated with the visual analog scale.
pain level | It was evaluated once day of the procedure, after the breast biopsy procedure.
  Pain felt during the breast biopsy was evaluated with the visual analog scale.
Satisfaction level with the procedure | It was evaluated once day of the procedure, after breast biopsy procedure.
  Satisfaction with the breast biopsy was evaluated.with the visual analog scale.
Satisfaction level with the education | It was evaluated once day of the procedure, after breast biopsy procedure.
  Satisfaction with the education was evaluated with the visual analog scale.
change readiness level | It was evaluated day of the procedure, just before the procedure.
  patients' level of readiness for the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No